CLINICAL TRIAL: NCT05673954
Title: Glaucoma Assessment Via Reading Ability Using Logarithmic Chinese Reading Acuity Chart
Brief Title: Glaucoma Assessment Via Reading Ability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2022800
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with primary open angle glaucoma
  Interventions: Diagnostic Test: C-Read test
- Control group: Healthy people
  Interventions: Diagnostic Test: C-Read test

INTERVENTIONS:
Diagnostic Test: C-Read test — C-Read is a reliable and valid clinical tool for quantitatively testing the reading ability of readers of simplified Chinese characters.

SUMMARY:
To explore a quantitative glaucoma evaluation tool of glaucoma through the dynamic evaluation of reading ability based on logarithmic Chinese reading acuity chart (C-READ), and investigate its feasibility.

DETAILED DESCRIPTION:
Glaucoma is the most common cause of irreversible blindness in the world, and it's marked by the gradual loss of retinal ganglion cells and their optic nerve fibres. Early detection and treatment can successfully prevent the disease's development and prevent blindness. Glaucoma sufferers' near visual qualities, particularly their ability to read, might be compromised. Patients can, however, regain some comfortable reading capacity following glaucoma therapy. The logarithmic Chinese reading acuity chart (C-READ) can be beneficial as a tool for functional vision evaluation, and there is rising clinical interest in this well-standardized, calibrated reading chart. Reading chart standards that allow for equal assessment of reading factors such as acuity and speed are currently lacking. The C-READ approach as a judge of glaucoma patients' status lacks theoretical support, and functional visual evaluation tools are still in their infancy. Therefore, we want to complete these tasks: 1) develop a dynamic analytic system and improve the evaluation criteria for the C-READ testing procedure; 2) confirm the usefulness of C-READ for early glaucoma screening through clinical studies. C-READ will provide a reliable and cost-effective screening technique that is convenient, affordable, and noninvasive.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma in at least 1 eye or labelled as a glaucoma suspect by a glaucoma specialist
* Age ≥18 years old
* with open angles on gonioscopy
* best-corrected visual acuity ≥0.5
* spherical refraction within ±5.0 diopters (D), and/or cylinder correction within 3.0 D

Exclusion Criteria:

* eyes with any evidence of physical abnormality of the iris or pupils on slit-lamp examination
* eyes with a history of trauma or inflammation
* undergone an intraocular surgery or laser within the previous 6 months/except uncomplicated cataract surgery
* using systemic or topical medications that could affect pupil responses, including pilocarpine or atropine
* presence of any media opacities that prevented good quality OCT or fundus images
* presence of any retinal or neurological disease other than glaucoma
* abnormal ocular motility that prevents binocular fixation (eg, nystagmus, strabismus)
* with severe systemic diseases or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who were diagnosed as primary open angle glaucoma in the Eye Center of the Third Hospital of Beijing Medical University from January 2023 to December 2023 will be included. At the same time, healthy people will be included as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
The Relationship between Reading Ability and C-READ Test Results | January 2023 to December 2023
  The Relationship between Reading Ability and C-READ Test Results